CLINICAL TRIAL: NCT02178618
Title: A Randomized Trial of Partially Covered Versus Uncovered Self Expandable Metal Stents for the Palliation of Malignant Distal Biliary Stricture
Brief Title: Partially Covered and Uncovered Metal Stent for Malignant Distal Biliary Stricture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jin Hong Kim, Professor, Ajou University School of Medicine
Other Study IDs: AJIRB-DEV-DE3-14-001
Record Dates: First submitted 2014-06-25; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Malignant Distal Biliary Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Partially covered biliary self expandable metal stent (Active Comparator)
  Interventions: Device: Deployment of Partially covered biliary self expandable metal stent
- Uncovered biliary self expandable metal stent (Active Comparator)
  Interventions: Device: Deployment of uncovered biliary self expandable metal stent

INTERVENTIONS:
Device: Deployment of Partially covered biliary self expandable metal stent
  Arms: Partially covered biliary self expandable metal stent
Device: Deployment of uncovered biliary self expandable metal stent
  Arms: Uncovered biliary self expandable metal stent

SUMMARY:
Endoscopic retrograde biliary drainage with a self-expandable metal stent (SEMS) has been used as a principle palliative method of distal biliary obstruction in patients with pancreaticobiliary cancers. With potentially curative surgical resection being impossible, the maintenance of successful biliary drainage through patent stent has been regarded as the key to improve the quality of life and survival of patient, because it could prevent biliary infection or liver failure, and give patients opportunities for anti-cancer chemotherapy and/or radiotherapy.

Although SEMSs have been reported to be superior to large bore plastic stents in terms of stent patency, they still have some controversial issues to resolve in relation to stent dysfunction and adverse event. It has been widely accepted that covered SEMSs designed to overcome the stent failure of uncovered SEMSs related to tumor ingrowth, have significant higher rate of stent migration as well as tumor overgrowth. Therefore covered SEMSs did not show the clear clinical excellence in the cumulative stent patency over uncovered SEMSs, despite some clinical results of randomized trials favor to covered SEMSs.

From the perspective of adverse events such as pancreatitis and cholecystitis, conflicting results have been produced. It was initially assumed that covered SEMSs could cause the higher incidence of pancreatitis and cholecystitis attributed to occlusion of pancreatic duct and cystic duct by covering materials. However, no significant difference was found with regard to the incidence of pancreatitis and cholecystitis between covered and uncovered SEMSs in several randomized trials and meta-analysis.

The aim of the current study is to compare the cumulative stent patency of partially covered and uncovered SEMS as a primary objective, and investigate overall patient survival, stent dysfunction-free patient survival, and incidence of adverse events including stent dysfunction as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

1. > 20 years
2. malignant biliary obstruction, 2 cm distal to hilum
3. unsuitable for curative surgical resection owing to metastasis, locally advanced stage, high operation risk, or patient's refusal
4. expected survival > 4 months based on Karnofsky performance score.

Exclusion Criteria:

1. history of biliary surgery except cholecystectomy
2. history of SEMS placement
3. coagulopathy (INR>1.5, Platelet<50000)
4. duodenal stricture

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Cumulative stent patency | From the date of randomization until the date of first documented stent dysfunction, assessed upto 12 months

SECONDARY OUTCOMES:
Overall patient survival | From the date of randomization until the date of death from any cause, assessed upto 12 months
Stent dysfunction free-patient survival | From the date of randomization until the date of first documented stent dysfunction or the date of death from any cause, whichever came first, assessed up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, Gyeong Gi Do, South Korea